CLINICAL TRIAL: NCT06344767
Title: Positive Estrogen Receptor (ER) Expression Assessed by 18F-fluoroestradiol Positron Emission Tomography/Computed Tomography (18F-FES PET/CT) in the Metastatic Breast Cancer (MBC) with ER- Negative Primary Tumor
Brief Title: Positive ER Expression Assessed by 18F-FES PET/CT in the MBC with ER-negative Primary Tumor
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-27
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FES positive in MBC: Patients who did not present with any ER-positive lesions in primary cancer were characterized as with any positive ER expression in the metastatic stage

SUMMARY:
To investigate the treatment pattern and efficacy of patients with negative primary ER lesion but positive ER expression in MBC using a novel convenient way of 18F-fluoroestradiol positron emission tomography/computed tomography (18F-FES PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer (according to International Classification of Diseases 10th Revision) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a nonmetastatic stage.
* MBC patients who underwent 18F-FES PET/CT at the Fudan University Shanghai Cancer Center between 2012 and 2023
* Patients diagnosed with primary ER-negative tumor and who were yet to receive any systemic therapy during the advanced stage

Exclusion Criteria:

Patients with incomplete medical records and those diagnosed with secondary primary tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MBC patients with ER-negative primary tumor who detected positive ER expression in metastatic disease using 18F-FES PET/CT at the Fudan University Shanghai Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- China,Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided